CLINICAL TRIAL: NCT03907553
Title: Aging of Hematopoietic Stem Cells - Molecular Architecture of Marrow Dysplasia and Clinical Contribution of Ineffective Hematopoiesis to Frailty in the Elderly
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Other Study IDs: CARIPLO 2016
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Anemia; Clonal Hematopoiesis
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health and Anemia: individuals belonging to the "Health and Anemia'' prospective population-based observational study (2003-2013) of all elderly residents (>65 years) in the municipality of Biella
  Interventions: Diagnostic Test: targeted genome sequencing
- Monzino: individuals belonging to the "Monzino Over 80 trial"
  Interventions: Diagnostic Test: targeted genome sequencing

INTERVENTIONS:
Diagnostic Test: targeted genome sequencing

SUMMARY:
The prevalence and incidence of anemia tend to increase with advancing age. Relatively low hemoglobin concentrations are a common laboratory finding in the elderly, for the most part judged by physicians as a sign without clinical relevance or as a marker of an underlying chronic disease having no independent influence on health.

In recent years several studies have started to challenge the widespread and self-perpetuating perception of anemia as an innocent bystander, reporting worse cognitive and quality of life outcomes and increased risk of hospitalization and mortality in the general population. Focusing on elderly people, anemia has a clear association with the phenotypic features of frailty syndrome affecting 3-5% of individuals of 65-70 years of age and, more importantly 30% of those aged 85 years or older.

Among frail older adults, anemia is a powerful prognostic factor for the development of frailty-related problems such as muscle weakness, reduced performance, falls, and mortality. Nutrient deficiency, chronic inflammation and renal insufficiency account for the large majority of cases of anemia in the elderly, while underlying cause remained unexplained in 25% of the cases. Preliminary evidence indicates that a significant proportion of ''unexplained anemia'' may account for myelodysplasia(MDS). MDS is a condition typically occurring in elderly people, characterized by clonal proliferation of hematopoietic stem cells (HSC), which partly retain their capacity to differentiate and maturate, but do so in an inefficient manner (ineffective hematopoiesis). Anemia represents the most important prognostic factor in MDS. With time a portion of patients evolve into overt myeloid malignancy (i.e., acute leukemia).

Somatic mutations occur in the genomes of healthy HSC at a low, but detectable frequency during normal DNA replication. Although most mutations are rapidly corrected by DNA repair mechanisms, those that persist are propagated during HSC self-renewal. Some evidence suggest that these early driver mutations dictate future trajectories of evolution with distinct clinical phenotypes. There has been much excitement in the research community about the translational opportunities offered by genome sequencing, possibly leading to the identification of specific types of mutational processes of how genome interact with environmental factors in determining clinical conditions associated with aging and to the implementation of a personalized molecular diagnosis and treatment for every patient. In this translational research project, using an integrated genomic analysis based on next generation sequencing (NGS) technologies,the investigators plan to dissect the genomic architecture of MDS, significantly contributing to many features of frailty and to individual vulnerability. The investigators will perform mutation analysis of candidate genes in a large and well characterized cohort of individuals belonging to the "Health and Anemia'' study. "Health and Anemia" is a prospective population-based observational study (2003-2013) of all elderly residents in the municipality of Biella, Piedmont, a town in the north-west of Italy. Hematological parameters together with data on cognition and functional status, mood and quality of life, fatigue, hospitalization and mortality were collected for all patients. Moreover, complete information on the development of hematological malignancies was provided by local tumor registry up to 2018. The investigators aim to identify genes associated with the induction of clonal hematopoiesis in elderly people, and then to correlate somatic mutations with clinical/hematological features and progression into MDS and/or overt leukemia. Moreover, The investigators will genotype single-cell-derived hematopoietic colonies from CD34+ compartments (hematopoietic stem cells, multipotent progenitors, common myeloid progenitors, and granulocyte progenitors) in order to clarify the clonal architecture of marrow dysplasia in HSC, the dynamics of clonal establishment and expansion during hematopoietic differentiation, and their relationship with the disease phenotype and evolution. Finally, by analysing clinical data from "Health and Anemia study" the investigators will investigate the clinical contribution of myelodysplasia-related anemia to the development of frailty syndrome and its clinical sequela. The definition of molecular architecture of marrow dysplasia would allow us to improve the current diagnosis and classification of anemia in the elderly and the assessment of individual patient's risk of disease associated morbidity/mortality. Finally, in patients with marrow dysplasia, gene sequencing is expected to predict the vulnerability of a particular genotype to specific treatment, thus providing a basis for optimizing at individual level timing and modality of therapeutic intervention. The study population of the MOnzino 80-plus study will be used as validation cohort.

ELIGIBILITY:
Health & Anemia Trial population

Inclusion Criteria:

* 65 years or older
* residence in the town of Biella, Italy
* consence fo biobanking

Exclusion Criteria:

No exclusion criteria other than age, residence and lack of a biobanked sample

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 4280 subjects with a biobanked blood sample available for genetic analysys out of the 8740 subjects enrolled in the Health & Anemia Trial.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2003-07 (Actual); Primary Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
genotype-phenotype correlation | 2016-2019
  genes associated with the induction of clonal hematopoiesis in elderly people, and then to correlate somatic mutations with clinical/hematological features and progression into MDS and/or overt leukemia

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guralnik JM, Eisenstaedt RS, Ferrucci L, Klein HG, Woodman RC. Prevalence of anemia in persons 65 years and older in the United States: evidence for a high rate of unexplained anemia. Blood. 2004 Oct 15;104(8):2263-8. doi: 10.1182/blood-2004-05-1812. Epub 2004 Jul 6. PMID 15238427
- [Background] Riva E, Tettamanti M, Mosconi P, Apolone G, Gandini F, Nobili A, Tallone MV, Detoma P, Giacomin A, Clerico M, Tempia P, Guala A, Fasolo G, Lucca U. Association of mild anemia with hospitalization and mortality in the elderly: the Health and Anemia population-based study. Haematologica. 2009 Jan;94(1):22-8. doi: 10.3324/haematol.13449. Epub 2008 Nov 10. PMID 19001283
- [Background] Rohrig G. Anemia in the frail, elderly patient. Clin Interv Aging. 2016 Mar 17;11:319-26. doi: 10.2147/CIA.S90727. eCollection 2016. PMID 27051279
- [Background] Juarez-Cedillo T, Basurto-Acevedo L, Vega-Garcia S, Manuel-Apolinar L, Cruz-Tesoro E, Rodriguez-Perez JM, Garcia-Hernandez N, Perez-Hernandez N, Fragoso JM. Prevalence of anemia and its impact on the state of frailty in elderly people living in the community: SADEM study. Ann Hematol. 2014 Dec;93(12):2057-62. doi: 10.1007/s00277-014-2155-4. Epub 2014 Jul 10. PMID 25005679
- [Background] Cazzola M, Malcovati L. Myelodysplastic syndromes--coping with ineffective hematopoiesis. N Engl J Med. 2005 Feb 10;352(6):536-8. doi: 10.1056/NEJMp048266. No abstract available. PMID 15703418
- [Background] Genovese G, Kahler AK, Handsaker RE, Lindberg J, Rose SA, Bakhoum SF, Chambert K, Mick E, Neale BM, Fromer M, Purcell SM, Svantesson O, Landen M, Hoglund M, Lehmann S, Gabriel SB, Moran JL, Lander ES, Sullivan PF, Sklar P, Gronberg H, Hultman CM, McCarroll SA. Clonal hematopoiesis and blood-cancer risk inferred from blood DNA sequence. N Engl J Med. 2014 Dec 25;371(26):2477-87. doi: 10.1056/NEJMoa1409405. Epub 2014 Nov 26. PMID 25426838
- [Background] Jaiswal S, Fontanillas P, Flannick J, Manning A, Grauman PV, Mar BG, Lindsley RC, Mermel CH, Burtt N, Chavez A, Higgins JM, Moltchanov V, Kuo FC, Kluk MJ, Henderson B, Kinnunen L, Koistinen HA, Ladenvall C, Getz G, Correa A, Banahan BF, Gabriel S, Kathiresan S, Stringham HM, McCarthy MI, Boehnke M, Tuomilehto J, Haiman C, Groop L, Atzmon G, Wilson JG, Neuberg D, Altshuler D, Ebert BL. Age-related clonal hematopoiesis associated with adverse outcomes. N Engl J Med. 2014 Dec 25;371(26):2488-98. doi: 10.1056/NEJMoa1408617. Epub 2014 Nov 26. PMID 25426837
- [Background] Papaemmanuil E, Gerstung M, Malcovati L, Tauro S, Gundem G, Van Loo P, Yoon CJ, Ellis P, Wedge DC, Pellagatti A, Shlien A, Groves MJ, Forbes SA, Raine K, Hinton J, Mudie LJ, McLaren S, Hardy C, Latimer C, Della Porta MG, O'Meara S, Ambaglio I, Galli A, Butler AP, Walldin G, Teague JW, Quek L, Sternberg A, Gambacorti-Passerini C, Cross NC, Green AR, Boultwood J, Vyas P, Hellstrom-Lindberg E, Bowen D, Cazzola M, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Clinical and biological implications of driver mutations in myelodysplastic syndromes. Blood. 2013 Nov 21;122(22):3616-27; quiz 3699. doi: 10.1182/blood-2013-08-518886. Epub 2013 Sep 12. PMID 24030381
- [Background] Cazzola M, Della Porta MG, Malcovati L. The genetic basis of myelodysplasia and its clinical relevance. Blood. 2013 Dec 12;122(25):4021-34. doi: 10.1182/blood-2013-09-381665. Epub 2013 Oct 17. PMID 24136165
- [Background] Ades L, Itzykson R, Fenaux P. Myelodysplastic syndromes. Lancet. 2014 Jun 28;383(9936):2239-52. doi: 10.1016/S0140-6736(13)61901-7. Epub 2014 Mar 21. PMID 24656536
- [Background] Malcovati L, Porta MG, Pascutto C, Invernizzi R, Boni M, Travaglino E, Passamonti F, Arcaini L, Maffioli M, Bernasconi P, Lazzarino M, Cazzola M. Prognostic factors and life expectancy in myelodysplastic syndromes classified according to WHO criteria: a basis for clinical decision making. J Clin Oncol. 2005 Oct 20;23(30):7594-603. doi: 10.1200/JCO.2005.01.7038. Epub 2005 Sep 26. PMID 16186598
- [Background] Malcovati L, Della Porta MG, Cazzola M. Predicting survival and leukemic evolution in patients with myelodysplastic syndrome. Haematologica. 2006 Dec;91(12):1588-90. No abstract available. PMID 17145593
- [Background] Della Porta MG, Travaglino E, Boveri E, Ponzoni M, Malcovati L, Papaemmanuil E, Rigolin GM, Pascutto C, Croci G, Gianelli U, Milani R, Ambaglio I, Elena C, Ubezio M, Da Via' MC, Bono E, Pietra D, Quaglia F, Bastia R, Ferretti V, Cuneo A, Morra E, Campbell PJ, Orazi A, Invernizzi R, Cazzola M; Rete Ematologica Lombarda (REL) Clinical Network. Minimal morphological criteria for defining bone marrow dysplasia: a basis for clinical implementation of WHO classification of myelodysplastic syndromes. Leukemia. 2015 Jan;29(1):66-75. doi: 10.1038/leu.2014.161. Epub 2014 May 20. PMID 24935723
- [Background] Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellstrom-Lindberg E, Tefferi A, Bloomfield CD. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. Blood. 2009 Jul 30;114(5):937-51. doi: 10.1182/blood-2009-03-209262. Epub 2009 Apr 8. PMID 19357394
- [Background] Snoeck HW. Aging of the hematopoietic system. Curr Opin Hematol. 2013 Jul;20(4):355-61. doi: 10.1097/MOH.0b013e3283623c77. PMID 23739721
- [Background] Yoshizato T, Dumitriu B, Hosokawa K, Makishima H, Yoshida K, Townsley D, Sato-Otsubo A, Sato Y, Liu D, Suzuki H, Wu CO, Shiraishi Y, Clemente MJ, Kataoka K, Shiozawa Y, Okuno Y, Chiba K, Tanaka H, Nagata Y, Katagiri T, Kon A, Sanada M, Scheinberg P, Miyano S, Maciejewski JP, Nakao S, Young NS, Ogawa S. Somatic Mutations and Clonal Hematopoiesis in Aplastic Anemia. N Engl J Med. 2015 Jul 2;373(1):35-47. doi: 10.1056/NEJMoa1414799. PMID 26132940
- [Background] Xie M, Lu C, Wang J, McLellan MD, Johnson KJ, Wendl MC, McMichael JF, Schmidt HK, Yellapantula V, Miller CA, Ozenberger BA, Welch JS, Link DC, Walter MJ, Mardis ER, Dipersio JF, Chen F, Wilson RK, Ley TJ, Ding L. Age-related mutations associated with clonal hematopoietic expansion and malignancies. Nat Med. 2014 Dec;20(12):1472-8. doi: 10.1038/nm.3733. Epub 2014 Oct 19. PMID 25326804
- [Background] Steensma DP, Bejar R, Jaiswal S, Lindsley RC, Sekeres MA, Hasserjian RP, Ebert BL. Clonal hematopoiesis of indeterminate potential and its distinction from myelodysplastic syndromes. Blood. 2015 Jul 2;126(1):9-16. doi: 10.1182/blood-2015-03-631747. Epub 2015 Apr 30. PMID 25931582
- [Background] Busque L, Patel JP, Figueroa ME, Vasanthakumar A, Provost S, Hamilou Z, Mollica L, Li J, Viale A, Heguy A, Hassimi M, Socci N, Bhatt PK, Gonen M, Mason CE, Melnick A, Godley LA, Brennan CW, Abdel-Wahab O, Levine RL. Recurrent somatic TET2 mutations in normal elderly individuals with clonal hematopoiesis. Nat Genet. 2012 Nov;44(11):1179-81. doi: 10.1038/ng.2413. Epub 2012 Sep 23. PMID 23001125
- [Background] Woll PS, Kjallquist U, Chowdhury O, Doolittle H, Wedge DC, Thongjuea S, Erlandsson R, Ngara M, Anderson K, Deng Q, Mead AJ, Stenson L, Giustacchini A, Duarte S, Giannoulatou E, Taylor S, Karimi M, Scharenberg C, Mortera-Blanco T, Macaulay IC, Clark SA, Dybedal I, Josefsen D, Fenaux P, Hokland P, Holm MS, Cazzola M, Malcovati L, Tauro S, Bowen D, Boultwood J, Pellagatti A, Pimanda JE, Unnikrishnan A, Vyas P, Gohring G, Schlegelberger B, Tobiasson M, Kvalheim G, Constantinescu SN, Nerlov C, Nilsson L, Campbell PJ, Sandberg R, Papaemmanuil E, Hellstrom-Lindberg E, Linnarsson S, Jacobsen SE. Myelodysplastic syndromes are propagated by rare and distinct human cancer stem cells in vivo. Cancer Cell. 2014 Jun 16;25(6):794-808. doi: 10.1016/j.ccr.2014.03.036. Epub 2014 May 15. PMID 24835589
- [Background] Ebert BL, Pretz J, Bosco J, Chang CY, Tamayo P, Galili N, Raza A, Root DE, Attar E, Ellis SR, Golub TR. Identification of RPS14 as a 5q- syndrome gene by RNA interference screen. Nature. 2008 Jan 17;451(7176):335-9. doi: 10.1038/nature06494. PMID 18202658
- [Background] Papaemmanuil E, Cazzola M, Boultwood J, Malcovati L, Vyas P, Bowen D, Pellagatti A, Wainscoat JS, Hellstrom-Lindberg E, Gambacorti-Passerini C, Godfrey AL, Rapado I, Cvejic A, Rance R, McGee C, Ellis P, Mudie LJ, Stephens PJ, McLaren S, Massie CE, Tarpey PS, Varela I, Nik-Zainal S, Davies HR, Shlien A, Jones D, Raine K, Hinton J, Butler AP, Teague JW, Baxter EJ, Score J, Galli A, Della Porta MG, Travaglino E, Groves M, Tauro S, Munshi NC, Anderson KC, El-Naggar A, Fischer A, Mustonen V, Warren AJ, Cross NC, Green AR, Futreal PA, Stratton MR, Campbell PJ; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium. Somatic SF3B1 mutation in myelodysplasia with ring sideroblasts. N Engl J Med. 2011 Oct 13;365(15):1384-95. doi: 10.1056/NEJMoa1103283. Epub 2011 Sep 26. PMID 21995386
- [Background] Yoshida K, Sanada M, Shiraishi Y, Nowak D, Nagata Y, Yamamoto R, Sato Y, Sato-Otsubo A, Kon A, Nagasaki M, Chalkidis G, Suzuki Y, Shiosaka M, Kawahata R, Yamaguchi T, Otsu M, Obara N, Sakata-Yanagimoto M, Ishiyama K, Mori H, Nolte F, Hofmann WK, Miyawaki S, Sugano S, Haferlach C, Koeffler HP, Shih LY, Haferlach T, Chiba S, Nakauchi H, Miyano S, Ogawa S. Frequent pathway mutations of splicing machinery in myelodysplasia. Nature. 2011 Sep 11;478(7367):64-9. doi: 10.1038/nature10496. PMID 21909114
- [Background] Malcovati L, Papaemmanuil E, Bowen DT, Boultwood J, Della Porta MG, Pascutto C, Travaglino E, Groves MJ, Godfrey AL, Ambaglio I, Galli A, Da Via MC, Conte S, Tauro S, Keenan N, Hyslop A, Hinton J, Mudie LJ, Wainscoat JS, Futreal PA, Stratton MR, Campbell PJ, Hellstrom-Lindberg E, Cazzola M; Chronic Myeloid Disorders Working Group of the International Cancer Genome Consortium and of the Associazione Italiana per la Ricerca sul Cancro Gruppo Italiano Malattie Mieloproliferative. Clinical significance of SF3B1 mutations in myelodysplastic syndromes and myelodysplastic/myeloproliferative neoplasms. Blood. 2011 Dec 8;118(24):6239-46. doi: 10.1182/blood-2011-09-377275. Epub 2011 Oct 12. PMID 21998214
- [Background] Dolatshad H, Pellagatti A, Fernandez-Mercado M, Yip BH, Malcovati L, Attwood M, Przychodzen B, Sahgal N, Kanapin AA, Lockstone H, Scifo L, Vandenberghe P, Papaemmanuil E, Smith CW, Campbell PJ, Ogawa S, Maciejewski JP, Cazzola M, Savage KI, Boultwood J. Disruption of SF3B1 results in deregulated expression and splicing of key genes and pathways in myelodysplastic syndrome hematopoietic stem and progenitor cells. Leukemia. 2015 May;29(5):1092-103. doi: 10.1038/leu.2014.331. Epub 2014 Nov 27. PMID 25428262
- [Background] Bejar R, Stevenson K, Abdel-Wahab O, Galili N, Nilsson B, Garcia-Manero G, Kantarjian H, Raza A, Levine RL, Neuberg D, Ebert BL. Clinical effect of point mutations in myelodysplastic syndromes. N Engl J Med. 2011 Jun 30;364(26):2496-506. doi: 10.1056/NEJMoa1013343. PMID 21714648
- [Background] Malcovati L, Hellstrom-Lindberg E, Bowen D, Ades L, Cermak J, Del Canizo C, Della Porta MG, Fenaux P, Gattermann N, Germing U, Jansen JH, Mittelman M, Mufti G, Platzbecker U, Sanz GF, Selleslag D, Skov-Holm M, Stauder R, Symeonidis A, van de Loosdrecht AA, de Witte T, Cazzola M; European Leukemia Net. Diagnosis and treatment of primary myelodysplastic syndromes in adults: recommendations from the European LeukemiaNet. Blood. 2013 Oct 24;122(17):2943-64. doi: 10.1182/blood-2013-03-492884. Epub 2013 Aug 26. PMID 23980065
- [Background] Greenberg PL, Tuechler H, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres M, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D. Revised international prognostic scoring system for myelodysplastic syndromes. Blood. 2012 Sep 20;120(12):2454-65. doi: 10.1182/blood-2012-03-420489. Epub 2012 Jun 27. PMID 22740453
- [Background] Della Porta MG, Tuechler H, Malcovati L, Schanz J, Sanz G, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Levis A, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Krieger O, Luebbert M, Maciejewski J, Magalhaes SM, Miyazaki Y, Pfeilstocker M, Sekeres MA, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D, Greenberg PL, Cazzola M. Validation of WHO classification-based Prognostic Scoring System (WPSS) for myelodysplastic syndromes and comparison with the revised International Prognostic Scoring System (IPSS-R). A study of the International Working Group for Prognosis in Myelodysplasia (IWG-PM). Leukemia. 2015 Jul;29(7):1502-13. doi: 10.1038/leu.2015.55. Epub 2015 Feb 27. PMID 25721895
- [Background] Schneider RK, Schenone M, Ferreira MV, Kramann R, Joyce CE, Hartigan C, Beier F, Brummendorf TH, Germing U, Platzbecker U, Busche G, Knuchel R, Chen MC, Waters CS, Chen E, Chu LP, Novina CD, Lindsley RC, Carr SA, Ebert BL. Rps14 haploinsufficiency causes a block in erythroid differentiation mediated by S100A8 and S100A9. Nat Med. 2016 Mar;22(3):288-97. doi: 10.1038/nm.4047. Epub 2016 Feb 15. PMID 26878232
- [Background] Itzykson R, Kosmider O, Cluzeau T, Mansat-De Mas V, Dreyfus F, Beyne-Rauzy O, Quesnel B, Vey N, Gelsi-Boyer V, Raynaud S, Preudhomme C, Ades L, Fenaux P, Fontenay M; Groupe Francophone des Myelodysplasies (GFM). Impact of TET2 mutations on response rate to azacitidine in myelodysplastic syndromes and low blast count acute myeloid leukemias. Leukemia. 2011 Jul;25(7):1147-52. doi: 10.1038/leu.2011.71. Epub 2011 Apr 15. PMID 21494260
- [Background] Itzykson R, Thepot S, Quesnel B, Dreyfus F, Beyne-Rauzy O, Turlure P, Vey N, Recher C, Dartigeas C, Legros L, Delaunay J, Salanoubat C, Visanica S, Stamatoullas A, Isnard F, Marfaing-Koka A, de Botton S, Chelghoum Y, Taksin AL, Plantier I, Ame S, Boehrer S, Gardin C, Beach CL, Ades L, Fenaux P; Groupe Francophone des Myelodysplasies(GFM). Prognostic factors for response and overall survival in 282 patients with higher-risk myelodysplastic syndromes treated with azacitidine. Blood. 2011 Jan 13;117(2):403-11. doi: 10.1182/blood-2010-06-289280. Epub 2010 Oct 12. PMID 20940414
- [Background] Blank U, Karlsson S. TGF-beta signaling in the control of hematopoietic stem cells. Blood. 2015 Jun 4;125(23):3542-50. doi: 10.1182/blood-2014-12-618090. Epub 2015 Apr 1. PMID 25833962
- [Background] Penninx BW, Pahor M, Cesari M, Corsi AM, Woodman RC, Bandinelli S, Guralnik JM, Ferrucci L. Anemia is associated with disability and decreased physical performance and muscle strength in the elderly. J Am Geriatr Soc. 2004 May;52(5):719-24. doi: 10.1111/j.1532-5415.2004.52208.x. PMID 15086651
- [Background] Penninx BW, Guralnik JM, Onder G, Ferrucci L, Wallace RB, Pahor M. Anemia and decline in physical performance among older persons. Am J Med. 2003 Aug 1;115(2):104-10. doi: 10.1016/s0002-9343(03)00263-8. PMID 12893395
- [Background] Cesari M, Penninx BW, Lauretani F, Russo CR, Carter C, Bandinelli S, Atkinson H, Onder G, Pahor M, Ferrucci L. Hemoglobin levels and skeletal muscle: results from the InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):249-54. doi: 10.1093/gerona/59.3.m249. PMID 15031309
- [Background] Ezekowitz JA, McAlister FA, Armstrong PW. Anemia is common in heart failure and is associated with poor outcomes: insights from a cohort of 12 065 patients with new-onset heart failure. Circulation. 2003 Jan 21;107(2):223-5. doi: 10.1161/01.cir.0000052622.51963.fc. PMID 12538418
- [Background] Hayashi T, Suzuki A, Shoji T, Togawa M, Okada N, Tsubakihara Y, Imai E, Hori M. Cardiovascular effect of normalizing the hematocrit level during erythropoietin therapy in predialysis patients with chronic renal failure. Am J Kidney Dis. 2000 Feb;35(2):250-6. doi: 10.1016/s0272-6386(00)70334-9. PMID 10676724
- [Background] Kim DH, Schneeweiss S. Measuring frailty using claims data for pharmacoepidemiologic studies of mortality in older adults: evidence and recommendations. Pharmacoepidemiol Drug Saf. 2014 Sep;23(9):891-901. doi: 10.1002/pds.3674. Epub 2014 Jun 24. PMID 24962929
- [Background] Artz AS. Anemia and the frail elderly. Semin Hematol. 2008 Oct;45(4):261-6. doi: 10.1053/j.seminhematol.2008.06.002. PMID 18809097
- [Background] Triscott JA, Dobbs BM, McKay RM, Babenko O, Triscott E. Prevalence and Types of Anemia and Associations with Functional Decline in Geriatric Inpatients. J Frailty Aging. 2015;4(1):7-12. doi: 10.14283/jfa.2015.35. PMID 27031910
- [Background] Ng TP, Feng L, Nyunt MS, Larbi A, Yap KB. Frailty in older persons: multisystem risk factors and the Frailty Risk Index (FRI). J Am Med Dir Assoc. 2014 Sep;15(9):635-42. doi: 10.1016/j.jamda.2014.03.008. Epub 2014 Apr 17. PMID 24746590
- [Background] Lucca U, Tettamanti M, Mosconi P, Apolone G, Gandini F, Nobili A, Tallone MV, Detoma P, Giacomin A, Clerico M, Tempia P, Guala A, Fasolo G, Riva E. Association of mild anemia with cognitive, functional, mood and quality of life outcomes in the elderly: the "Health and Anemia" study. PLoS One. 2008 Apr 2;3(4):e1920. doi: 10.1371/journal.pone.0001920. PMID 18382689
- [Background] Malcovati L, Karimi M, Papaemmanuil E, Ambaglio I, Jadersten M, Jansson M, Elena C, Galli A, Walldin G, Della Porta MG, Raaschou-Jensen K, Travaglino E, Kallenbach K, Pietra D, Ljungstrom V, Conte S, Boveri E, Invernizzi R, Rosenquist R, Campbell PJ, Cazzola M, Hellstrom Lindberg E. SF3B1 mutation identifies a distinct subset of myelodysplastic syndrome with ring sideroblasts. Blood. 2015 Jul 9;126(2):233-41. doi: 10.1182/blood-2015-03-633537. Epub 2015 May 8. PMID 25957392
- [Background] Malcovati L, Papaemmanuil E, Ambaglio I, Elena C, Galli A, Della Porta MG, Travaglino E, Pietra D, Pascutto C, Ubezio M, Bono E, Da Via MC, Brisci A, Bruno F, Cremonesi L, Ferrari M, Boveri E, Invernizzi R, Campbell PJ, Cazzola M. Driver somatic mutations identify distinct disease entities within myeloid neoplasms with myelodysplasia. Blood. 2014 Aug 28;124(9):1513-21. doi: 10.1182/blood-2014-03-560227. Epub 2014 Jun 26. PMID 24970933
- [Background] Shirai CL, Ley JN, White BS, Kim S, Tibbitts J, Shao J, Ndonwi M, Wadugu B, Duncavage EJ, Okeyo-Owuor T, Liu T, Griffith M, McGrath S, Magrini V, Fulton RS, Fronick C, O'Laughlin M, Graubert TA, Walter MJ. Mutant U2AF1 Expression Alters Hematopoiesis and Pre-mRNA Splicing In Vivo. Cancer Cell. 2015 May 11;27(5):631-43. doi: 10.1016/j.ccell.2015.04.008. PMID 25965570
- [Background] Kim E, Ilagan JO, Liang Y, Daubner GM, Lee SC, Ramakrishnan A, Li Y, Chung YR, Micol JB, Murphy ME, Cho H, Kim MK, Zebari AS, Aumann S, Park CY, Buonamici S, Smith PG, Deeg HJ, Lobry C, Aifantis I, Modis Y, Allain FH, Halene S, Bradley RK, Abdel-Wahab O. SRSF2 Mutations Contribute to Myelodysplasia by Mutant-Specific Effects on Exon Recognition. Cancer Cell. 2015 May 11;27(5):617-30. doi: 10.1016/j.ccell.2015.04.006. PMID 25965569
- [Background] Robusto M, Fang M, Asselta R, Castorina P, Previtali SC, Caccia S, Benzoni E, De Cristofaro R, Yu C, Cesarani A, Liu X, Li W, Primignani P, Ambrosetti U, Xu X, Duga S, Solda G. The expanding spectrum of PRPS1-associated phenotypes: three novel mutations segregating with X-linked hearing loss and mild peripheral neuropathy. Eur J Hum Genet. 2015 Jun;23(6):766-73. doi: 10.1038/ejhg.2014.168. Epub 2014 Sep 3. PMID 25182139
- [Background] Lucca U, Tettamanti M, Logroscino G, Tiraboschi P, Landi C, Sacco L, Garri M, Ammesso S, Bertinotti C, Biotti A, Gargantini E, Piedicorcia A, Nobili A, Pasina L, Franchi C, Djade CD, Riva E, Recchia A. Prevalence of dementia in the oldest old: the Monzino 80-plus population based study. Alzheimers Dement. 2015 Mar;11(3):258-70.e3. doi: 10.1016/j.jalz.2014.05.1750. Epub 2014 Aug 20. PMID 25150732
- [Background] Lucca U, Garri M, Recchia A, Logroscino G, Tiraboschi P, Franceschi M, Bertinotti C, Biotti A, Gargantini E, Maragna M, Nobili A, Pasina L, Franchi C, Riva E, Tettamanti M. A Population-based study of dementia in the oldest old: the Monzino 80-plus study. BMC Neurol. 2011 May 25;11:54. doi: 10.1186/1471-2377-11-54. PMID 21612585
- [Result] Tettamanti M, Lucca U, Gandini F, Recchia A, Mosconi P, Apolone G, Nobili A, Tallone MV, Detoma P, Giacomin A, Clerico M, Tempia P, Savoia L, Fasolo G, Ponchio L, Della Porta MG, Riva E. Prevalence, incidence and types of mild anemia in the elderly: the "Health and Anemia" population-based study. Haematologica. 2010 Nov;95(11):1849-56. doi: 10.3324/haematol.2010.023101. Epub 2010 Jun 9. PMID 20534701
- [Derived] Da Via MC, Lionetti M, Marella A, Matera A, Travaglino E, Signaroldi E, Galbussera AA, Lucca U, Mandelli S, Riva E, Tettamanti M, Pettine L, Pompa A, Baldini L, Neri A, Della Porta MG, Bolli N. MGUS and clonal hematopoiesis show unrelated clinical and biological trajectories in an older population cohort. Blood Adv. 2022 Nov 8;6(21):5702-5706. doi: 10.1182/bloodadvances.2021006498. PMID 35390146